CLINICAL TRIAL: NCT00099372
Title: Long-term Effectiveness of Abdominal Sacrocolpopexy for the Treatment of Pelvic Organ Prolapse: The Extended Colpopexy and Urinary Reduction Efforts (E-CARE) Study
Brief Title: Long-term Effectiveness of Abdominal Sacrocolpopexy for the Treatment of Pelvic Organ Prolapse
Acronym: E-CARE
Status: Terminated | Type: Observational
Why Stopped: resource and prioritization change as Network transition to a new funding cycle
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: University of Iowa (Other); Baylor College of Medicine (Other); Loyola University (Other); University of North Carolina, Chapel Hill (Other); Johns Hopkins University (Other); University of Pittsburgh (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PFD 001; U01HD41249; U01HD041249 (NIH); U10HD041268 (NIH); U10HD041248 (NIH); U10HD041250 (NIH); U10HD041261 (NIH); U10HD041263 (NIH); U10HD041269 (NIH); U10HD041267 (NIH)
Record Dates: First submitted 2004-12-10; First posted 2004-12-13 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2020-12

CONDITIONS: Prolapse; Urinary Incontinence
Keywords: sacrocolpopexy; abdominal sacrocolpopexy; surgical procedure, prolapse; pelvic organ prolapse; urinary incontinence; stress urinary incontinence
MeSH Terms: conditions — Prolapse; Urinary Incontinence; Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Abdominal Sacral Colpopexy with no Burch colposuspension: Participants had an Abdominal Sacral Colpopexy without Burch colposuspension for treatment of pelvic organ prolapse
- Abdominal Sacral Colpopexy with Burch Colposuspension: Participants had an Abdominal Sacral Colpopexy with Burch colposuspension for treatment of pelvic organ prolapse

SUMMARY:
The Colpopexy and Urinary Reduction Effort (CARE) trial is a research study designed to evaluate whether the addition of a second surgical procedure in addition to a procedure for female pelvic organ prolapse (POP) affects the rates of urinary incontinence. This study will follow women in the CARE study for 10 years from the time of the surgery to compare success and complication rates in the two groups. Recruitment into this study is open only to women that already participated in CARE. Recruitment into CARE is closed.

DETAILED DESCRIPTION:
The primary aims of this prospective cohort study are:

1. To determine the long-term (up to 10 years) anatomic success rate of sacrocolpopexy (defined as Stage 0 apical prolapse AND <= Stage 2 anterior and posterior prolapse AND no re-operation or pessary treatment for POP), and whether anatomic success differs between women who had vs. those who did not have concomitant Burch colposuspension at the time of sacrocolpopexy;
2. To determine whether there is a difference in long-term stress continence (by symptoms) between women who had vs. those who did not have concomitant Burch colposuspension at the time of sacrocolpopexy;
3. To determine whether there is a long-term difference between overall pelvic floor symptoms and pelvic-floor specific quality of life between women who had vs. those who did not have concomitant Burch colposuspension at the time of sacrocolpopexy.

ELIGIBILITY:
Inclusion Criteria:

* Women enrolled in CARE

Exclusion Criteria:

* Inability to provide informed consent.
* Subjects who, at the time of enrollment into E-CARE, are long-term residents of a skilled nursing facility (that is, residency is not limited to short-term rehabilitation).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who completed the CARE study
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2004-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Nygaard, MD, Study Chair — University of Utah
Locations (8):
- United States (8):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - USCD Medical Center, La Jolla, California
  - Kaiser Permanente, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Nygaard I, Brubaker L, Zyczynski HM, Cundiff G, Richter H, Gantz M, Fine P, Menefee S, Ridgeway B, Visco A, Warren LK, Zhang M, Meikle S. Long-term outcomes following abdominal sacrocolpopexy for pelvic organ prolapse. JAMA. 2013 May 15;309(19):2016-24. doi: 10.1001/jama.2013.4919. PMID 23677313

RESULTS

PARTICIPANT FLOW:
Period: Enrolled in Extended CARE Trial
Arm/Group | Abdominal Sacral Colpopexy With Burch Colposuspension | Abdominal Sacral Colpopexy With No Burch Colposuspension
Started | 104 | 111
Completed | 104 | 111
Not Completed | 0 | 0
Period: Followed up 5 Years After Index Surgery
Arm/Group | Abdominal Sacral Colpopexy With Burch Colposuspension | Abdominal Sacral Colpopexy With No Burch Colposuspension
Started | 104 | 111
Completed | 89 | 92
Not Completed | 15 | 19
Period: Followed up 7 Years After Index Surgery
Arm/Group | Abdominal Sacral Colpopexy With Burch Colposuspension | Abdominal Sacral Colpopexy With No Burch Colposuspension
Started | 89 | 92
Completed | 66 | 60
Not Completed | 23 | 32

BASELINE CHARACTERISTICS:
Groups:
- BURCH URETHROPEXY: Participants had an Abdominal Sacral Colpopexy with Burch colposuspension for treatment of pelvic organ prolapse
- NO URETHROPEXY: Participants had an Abdominal Sacral Colpopexy without Burch colposuspension for treatment of pelvic organ prolapse
- Total: Total of all reporting groups
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY | Total
Number analyzed (Participants) | 104 | 111 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.4) | 60.9 (10.5) | 61.9 (10)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 104 | 111 | 215
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4 | 9 | 13
  Other | 1 | 3 | 4
  White | 99 | 99 | 198
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1 | 7 | 8
  Not Hispanic | 103 | 104 | 207
Married or living as married [Count of Participants; unit: Participants]
  Missing | 1 | 0 | 1
  No | 23 | 31 | 54
  Yes | 80 | 80 | 160
Education level [Count of Participants; unit: Participants]
  College degree or higher | 53 | 63 | 116
  High school degree or equivalent | 36 | 44 | 80
  Less than High School | 15 | 4 | 19
Number of vaginal deliveries [Median (Full Range); unit: deliveries] | 3 [0 to 8] | 3 [1 to 8] | 3 [0 to 8]
Number of cesarean deliveries [Median (Full Range); unit: deliveries] | 0 [0 to 5] | 0 [0 to 2] | 0 [0 to 5]
Number of previous births [Median (Full Range); unit: births] | 3 [1 to 10] | 3 [1 to 8] | 3 [1 to 10]
Hysterectomy [Count of Participants; unit: Participants]
  Missing | 17 | 15 | 32
  No | 7 | 17 | 24
  Yes | 80 | 79 | 159
Prior SUI Surgery [Count of Participants; unit: Participants]
  No | 95 | 104 | 199
  Yes | 9 | 7 | 16
Prior POP Surgery [Count of Participants; unit: Participants]
  No | 56 | 75 | 131
  Yes | 48 | 36 | 84
Pelvic Organ Prolapse-Q stage [Count of Participants; unit: Participants] — The POP-Q assessment is a tool that measures the severity of prolapse. It measures nine points in the vagina with the hymen being the reference point. The distance to the reference point (in cm) is measured and the prolapse severity stage is calculated based on those measures. Higher stages indicate worse prolapse.
  Participants
    2 | 9 | 15 | 24
    3 | 75 | 78 | 153
    4 | 20 | 18 | 38
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (4) | 26.8 (4.8) | 26.7 (4.4)
BMI >= 30 (obesity) [Count of Participants; unit: Participants]
  No | 85 | 85 | 170
  Yes | 19 | 26 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic Failure
Description: Symptom of bulge on Pelvic Floor Distress Inventory, interval prolapse surgery, or pessary used after index surgery
Time Frame: 24 months
Population: This outcome is analyzed in randomized participants who completed the visit at this time point, or who were failures prior to the time point. Excluded from the analyses are prior dropouts who had not yet met the failure criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 104 | 111
Participants
  Failure | 15 | 16
  Non-failure | 89 | 95

2. Primary Outcome: Number of Participants With Symptomatic Failure
Description: Symptom of bulge on Pelvic Floor Distress Inventory, interval prolapse surgery, or pessary used after index surgery
Time Frame: 3 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- BURCH URETHROPEXY: Abdominal Sacral Colpopexy with Burch Colposuspension
- NO URETHROPEXY: Abdominal Sacral Colpopexy with No Burch Colposuspension
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 101 | 108
Participants
  Failure | 16 | 19
  Non-failure | 85 | 89

3. Primary Outcome: Number of Participants With Symptomatic Failure
Description: Symptom of bulge on Pelvic Floor Distress Inventory, interval prolapse surgery, or pessary used after index surgery
Time Frame: 4 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 94 | 103
Participants
  Failure | 19 | 20
  Non-failure | 75 | 83

4. Primary Outcome: Number of Participants With Symptomatic Failure
Description: Symptom of bulge on Pelvic Floor Distress Inventory, interval prolapse surgery, or pessary used after index surgery
Time Frame: 5 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 91 | 96
Participants
  Failure | 25 | 21
  Non-failure | 66 | 75

5. Primary Outcome: Number of Participants With Symptomatic Failure
Description: Symptom of bulge on Pelvic Floor Distress Inventory, interval prolapse surgery, or pessary used after index surgery
Time Frame: 6 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 86 | 90
Participants
  Failure | 27 | 21
  Non-failure | 59 | 69

6. Primary Outcome: Number of Participants With Symptomatic Failure
Description: Symptom of bulge on Pelvic Floor Distress Inventory, interval prolapse surgery, or pessary used after index surgery
Time Frame: 7 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 73 | 71
Participants
  Failure | 27 | 22
  Non-failure | 46 | 49

7. Primary Outcome: Number of Participants With Anatomic Failure (Original Definition)
Description: Reoperation or pessary for POP or POP-Q measurements as follows: Vaginal apex decends >= 2 cm, or the anterior or posterior vaginal wall decends >1 cm beyond the hymen
Time Frame: 24 months
Population: This outcome is analyzed in randomized participants who completed the visit at this time point, or who were failures prior to the time point. Excluded from the analyses are prior dropouts who had not yet met the failure criteria. The original and updated versions of anatomic failure could have different denominators for the same time point because a prior anatomic failure means the patient is assigned a failure in all subsequent visits regardless of whether the patient had completed the visits.
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 101 | 110
Participants
  Failure | 6 | 9
  Non-failure | 95 | 101

8. Primary Outcome: Number of Participants With Anatomic Failure (Original Definition)
Description: as for outcome 7
Time Frame: 3 year
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 84 | 90
Participants
  Failure | 9 | 10
  Non-failure | 75 | 80

9. Primary Outcome: Number of Participants With Anatomic Failure (Original Definition)
Description: as for outcome 7
Time Frame: 4 year
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 64 | 77
Participants
  Failure | 10 | 12
  Non-failure | 54 | 65

10. Primary Outcome: Number of Participants With Anatomic Failure (Original Definition)
Description: as for outcome 7
Time Frame: 5 year
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 58 | 69
Participants
  Failure | 12 | 13
  Non-failure | 46 | 56

11. Primary Outcome: Number of Participants With Anatomic Failure (Original Definition)
Description: as for outcome 7
Time Frame: 6 year
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 55 | 56
Participants
  Failure | 15 | 14
  Non-failure | 40 | 42

12. Primary Outcome: Number of Participants With Anatomic Failure (Original Definition)
Description: as for outcome 7
Time Frame: 7 year
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 44 | 46
Participants
  Failure | 15 | 14
  Non-failure | 29 | 32

13. Primary Outcome: Number of Participants With Anatomic Failure (Updated Definition)
Description: Reoperation or pessary for POP or POP-Q measurements as follows: Vaginal apex descends below the upper third of the vagina, or the anterior (Ba) or posterior (Bp) vaginal wall prolapses beyond the hymen
Time Frame: 24 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 101 | 110
Participants
  Failure | 5 | 8
  Non-failure | 96 | 102

14. Primary Outcome: Number of Participants With Anatomic Failure (Updated Definition)
Description: as for outcome 13
Time Frame: 3 year
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 84 | 91
Participants
  Failure | 8 | 10
  Non-failure | 76 | 81

15. Primary Outcome: Number of Participants With Anatomic Failure (Updated Definition)
Description: as for outcome 13
Time Frame: 4 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 64 | 79
Participants
  Failure | 10 | 12
  Non-failure | 54 | 67

16. Primary Outcome: Number of Participants With Anatomic Failure (Updated Definition)
Description: as for outcome 13
Time Frame: 5 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 56 | 71
Participants
  Failure | 14 | 12
  Non-failure | 42 | 59

17. Primary Outcome: Number of Participants With Anatomic Failure (Updated Definition)
Description: as for outcome 13
Time Frame: 6 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 54 | 59
Participants
  Failure | 18 | 13
  Non-failure | 36 | 46

18. Primary Outcome: Number of Participants With Anatomic Failure (Updated Definition)
Description: as for outcome 13
Time Frame: 7 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 45 | 49
Participants
  Failure | 18 | 13
  Non-failure | 27 | 36

19. Primary Outcome: Number of Participants With Composite Failure
Description: Anatomic failure (updated definition) or symptomatic failure
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 102 | 110
Participants
  Failure | 14 | 15
  Non-failure | 88 | 95

20. Primary Outcome: Number of Participants With Composite Failure
Description: Anatomic failure (updated definition) or symptomatic failure
Time Frame: 3 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 89 | 92
Participants
  Failure | 16 | 18
  Non-failure | 73 | 74

21. Primary Outcome: Number of Participants With Composite Failure
Description: Anatomic failure (updated definition) or symptomatic failure
Time Frame: 4 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 70 | 82
Participants
  Failure | 19 | 19
  Non-failure | 51 | 63

22. Primary Outcome: Number of Participants With Composite Failure
Description: Anatomic failure (updated definition) or symptomatic failure
Time Frame: 5 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 63 | 75
Participants
  Failure | 27 | 20
  Non-failure | 36 | 55

23. Primary Outcome: Number of Participants With Composite Failure
Description: Anatomic failure (updated definition) or symptomatic failure
Time Frame: 6 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 61 | 66
Participants
  Failure | 30 | 21
  Non-failure | 31 | 45

24. Primary Outcome: Number of Participants With Composite Failure
Description: Anatomic failure (updated definition) or symptomatic failure
Time Frame: 7 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 54 | 61
Participants
  Failure | 30 | 21
  Non-failure | 24 | 40

25. Primary Outcome: Number of Participants Considered as Failures For Urinary Incontinence Using the Incontinence Severity Index
Description: Failure is indicated by a score of 3 or greater on the Incontinence Severity Index (formerly called Hunskaar). The score is calculated as the product of the answers to two incontinence-related questions resulting in a range from 0 to 12 (higher scores indicating more severe symptoms). A score of 3 or greater corresponds to a severity classification of moderate, severe, or very severe.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 104 | 111
Participants
  Failure | 48 | 66
  Non-failure | 56 | 45

26. Primary Outcome: Number of Participants Considered as Failures For Urinary Incontinence Using the Incontinence Severity Index
Description: as for outcome 25
Time Frame: 3 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 101 | 109
Participants
  Failure | 52 | 70
  Non-failure | 49 | 39

27. Primary Outcome: Number of Participants Considered as Failures For Urinary Incontinence Using the Incontinence Severity Index
Description: as for outcome 25
Time Frame: 4 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 99 | 105
Participants
  Failure | 55 | 70
  Non-failure | 44 | 35

28. Primary Outcome: Number of Participants Considered as Failures For Urinary Incontinence Using the Incontinence Severity Index
Description: as for outcome 25
Time Frame: 5 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 98 | 104
Participants
  Failure | 58 | 72
  Non-failure | 40 | 32

29. Primary Outcome: Number of Participants Considered as Failures For Urinary Incontinence Using the Incontinence Severity Index
Description: as for outcome 25
Time Frame: 6 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 97 | 102
Participants
  Failure | 59 | 73
  Non-failure | 38 | 29

30. Primary Outcome: Number of Participants Considered as Failures For Urinary Incontinence Using the Incontinence Severity Index
Description: as for outcome 25
Time Frame: 7 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 91 | 92
Participants
  Failure | 62 | 73
  Non-failure | 29 | 19

31. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI) Prevention
Description: One or more SUI symptoms reported on the Pelvic Floor Distress Inventory, receipt of interval anti-incontinence surgery, or receipt of an urethral bulking agent injection for SUI
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 104 | 110
Participants
  Failure | 39 | 63
  Non-failure | 65 | 47

32. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI) Prevention
Description: as for outcome 31
Time Frame: 3 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 102 | 109
Participants
  Failure | 47 | 69
  Non-failure | 55 | 40

33. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI) Prevention
Description: as for outcome 31
Time Frame: 4 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 99 | 107
Participants
  Failure | 49 | 76
  Non-failure | 50 | 31

34. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI) Prevention
Description: as for outcome 31
Time Frame: 5 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 98 | 105
Participants
  Failure | 53 | 77
  Non-failure | 45 | 28

35. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI) Prevention
Description: as for outcome 31
Time Frame: 6 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 95 | 105
Participants
  Failure | 55 | 78
  Non-failure | 40 | 27

36. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI) Prevention
Description: as for outcome 31
Time Frame: 7 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 89 | 96
Participants
  Failure | 57 | 79
  Non-failure | 32 | 17

37. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI)
Description: One or more SUI symptoms reported on the Pelvic Floor Distress Inventory
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 104 | 110
Participants
  Failure | 39 | 63
  Non-failure | 65 | 47

38. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI)
Description: One or more SUI symptoms reported on the Pelvic Floor Distress Inventory
Time Frame: 3 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 102 | 109
Participants
  Failure | 47 | 68
  Non-failure | 55 | 41

39. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI)
Description: One or more SUI symptoms reported on the Pelvic Floor Distress Inventory
Time Frame: 4 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 99 | 107
Participants
  Failure | 49 | 75
  Non-failure | 50 | 32

40. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI)
Description: One or more SUI symptoms reported on the Pelvic Floor Distress Inventory
Time Frame: 5 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 98 | 105
Participants
  Failure | 53 | 76
  Non-failure | 45 | 29

41. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI)
Description: One or more SUI symptoms reported on the Pelvic Floor Distress Inventory
Time Frame: 6 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 95 | 105
Participants
  Failure | 55 | 78
  Non-failure | 40 | 27

42. Primary Outcome: Number of Participants With Stress Urinary Incontinence (SUI)
Description: One or more SUI symptoms reported on the Pelvic Floor Distress Inventory
Time Frame: 7 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BURCH URETHROPEXY | NO URETHROPEXY
Number analyzed (Participants) | 89 | 96
Participants
  Failure | 57 | 79
  Non-failure | 32 | 17

ADVERSE EVENTS:
Arm/Group | Abdominal Sacral Colpopexy With Burch Colposuspension | Abdominal Sacral Colpopexy With No Burch Colposuspension
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/111
Other Adverse Events (participants affected / at risk) | 12/104 | 15/111
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal Sacral Colpopexy With Burch Colposuspension (N=104) | Abdominal Sacral Colpopexy With No Burch Colposuspension (N=111)
Medical device site reaction (Surgical and medical procedures) | 11 (11) | 12 (12) — Mesh Erosion
Medical device site reaction (Surgical and medical procedures) | 1 (1) | 3 (3) — Suture Erosion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No